CLINICAL TRIAL: NCT04130542
Title: An Open Label, First in Human (FIH), Phase 1 Trial of LVGN6051 as Single Agent and in Combination With Keytruda (Pembrolizumab) in Advanced or Metastatic Malignancy
Brief Title: Phase 1 Trial of LVGN6051 as Single Agent and in Combination With Keytruda (Pembrolizumab) in Advanced or Metastatic Malignancy
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Lyvgen Biopharma Holdings Limited (Industry)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LVGN6051-101; MK-3475-A31/KEYNOTE-A31 (Other: Merck Sharp & Dohme LLC)
Record Dates: First submitted 2019-10-14; First posted 2019-10-17 (Actual); Last update posted 2024-10-31 (Actual); Status verified 2024-10

CONDITIONS: Cancer
Keywords: Lyvgen; MK-3475; Pembrolizumab; Keytruda
MeSH Terms: conditions — Neoplasms | interventions — pembrolizumab

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- LVGN6051 (Experimental): The dose escalation phase includes 10 dose levels of LVGN6051, and the highest dose is up to 10mg/kg. Route of administration is IV infusion, and the frequency of administration is once every 3 weeks (Q3W). one cycle is 3 weeks, and treatment can be up to 35 cycles if patients receive benefits.
  Interventions: Biological: LVGN6051; Biological: KEYTRUDA® (pembrolizumab)

INTERVENTIONS:
Biological: LVGN6051 — IV infusion once every 3 weeks (Q3W).
Biological: KEYTRUDA® (pembrolizumab) — IV infusion once every 3 weeks (Q3W).

SUMMARY:
LVGN6051 is a humanized monoclonal antibody that specifically binds to CD137, and acts as an agonist against CD137.

This first in human study of LVGN6051 is designed to establish the maximum tolerated dose (MTD) and/or the recommended dose for expansion (RDE) as well as the recommended Phase 2 dose(s) (RP2D) of LVGN6051, both as a single agent (monotherapy) and in combination with a fixed dose of anti-PD-1 antibody (Pembrolizumab/MK-3475) in the treatment of advanced or metastatic malignancy.

DETAILED DESCRIPTION:
This is an open-label, non-randomized, two-stage, FIH Phase 1 study, utilizing an accelerated dose escalation followed by a traditional 3 + 3 dose escalation algorithm to identify the MTD and/or RDE and RP2D of LVGN6051 as a single agent (monotherapy) and in combination with pembrolizumab (MK-3475). The first stage of the study is the dose escalation phase (i.e., Phase 1a). The second stage of the study is the dose expansion phase (i.e., Phase 1b). During the study, dose interruption(s) and/or delay(s) may be implemented based on toxicity. Dose modifications are not permitted. Intra-patient dose escalations will be allowed for the early dose cohorts (single-patient dose groups) in Phase 1a Part 1. Patients will be considered evaluable for safety and tolerability if they receive at least one dose of LVGN6051 or pembrolizumab (MK-3475) at the specified cohort dose. Patients in all parts of the trial will remain on therapy until confirmed disease progression or for 2 years, whichever occurs first. However, patients who are clinically unstable will discontinue following the initial assessment of disease progression.

ELIGIBILITY:
Inclusion Criteria:

* Males or females aged ≥ 18 years.
* Ability to understand and willingness to sign a written informed consent document.
* Patients must have a histologically or cytologically confirmed metastatic or unresectable malignancy.
* Estimated life expectancy, in the judgment of the Investigator, of at least 90 days.
* Adequate bone marrow, liver, and renal functions.
* Men and women of childbearing potential must agree to take highly effective contraceptive methods.
* Patients should recover from all reversible AEs of previous anticancer therapies to baseline.
* Patients infected with the HIV virus will be eligible if the disease is under control of effective therapy.

Exclusion Criteria:

* Receipt of systemic anticancer therapy including investigational agents or devices within 5 half-lives of the first dose of study treatment.
* Previous radiotherapy within 14 days of the first dose of study treatment.
* Known active CNS metastasis and/or carcinomatous meningitis.
* Has received a live-virus vaccine within 30 days.
* Has had a Grade ≥ 3 allergic reaction to treatment with a monoclonal antibody.
* Abnormality of QT interval or syndrome.
* Patients with history of Grade ≥ 3 immune-related AEs (irAEs) or irAE.
* Patients who are receiving an immunologically-based treatment for any reason.
* Treatment with systemic immune-stimulatory agents within 4 weeks prior to the first dose of study drug.
* Active or chronic autoimmune disease that has required systemic treatment in the past 2 years or who are receiving systemic therapy for an autoimmune or inflammatory disease.
* Has a clinically significant cardiac condition, including unstable angina, acute myocardial infarction within 6 months.
* Has an active infection requiring intravenous (i.v.) anti-infectives within 14 days before the first dose of study treatment.
* Current evidence or history of interstitial lung disease or active, noninfectious pneumonitis requiring treatment such as oral or intravenous glucocorticoids to assist with management.
* Female patients who are pregnant or breastfeeding.
* Any evidence of severe or uncontrolled systemic disease.
* Any other disease or clinically significant abnormality in laboratory parameters.
* Has previously had a stem cell or bone marrow or solid organ transplant.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 276 (Estimated)
Dates: Start 2019-10-31 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Safety/Tolerability | up to 24 months
  mEvaluate the safety and tolerability and determine the Maximum tolerated dose (MTD) and/or recommended dose for expansion (RDE) and recommended Phase 2 dose(s) (RP2D) of LVGN6051 administered as a single agent (monotherapy) and in combination with pembrolizumab, in adult patients with advanced malignancy.

CONTACTS AND LOCATIONS:
Locations (7):
- United States (7):
  - University of California Irvine Health, Orange, California
  - UCSF Helen Diller Family Comprehensive Cancer Center, San Francisco, California
  - Verdi Oncology Research, Lafayette, Indiana
  - The Johns Hopkins University, Baltimore, Maryland
  - Nebraska Cancer Specialist, Omaha, Nebraska
  - NYU Langone Health, New York, New York
  - MD Anderson Cancer Center, Houston, Texas